CLINICAL TRIAL: NCT00677443
Title: A Randomized Phase III Study of SOX vs. COX in Patients With Advanced Colorectal Cancer
Brief Title: Study of S-1 and Oxaliplatin (SOX) Versus Capecitabine and Oxaliplatin (COX) in Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: National Cancer Center, Korea (Other Government); Seoul National University Bundang Hospital (Other); Seoul National University Hospital (Other); Gachon University Gil Medical Center (Other); Yonsei University (Other); Asan Medical Center (Other); Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Young Suk Park, M.D.,Ph.D. Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-03-012
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Cancer
Keywords: metastatic colorectal cancer; S-1; Capecitabine; Oxaliplatin; non-inferiority study
MeSH Terms: conditions — Colorectal Neoplasms | interventions — S 1 (combination); Oxaliplatin; XELOX; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-1 and Oxaliplatin (Experimental): S-1 and Oxaliplatin
  S-1 : 80 mg/m2/day D1-14 Oxaliplatin : 130 mg/m2/day D1 Repeated every 3 weeks
  Interventions: Drug: S-1 & Oxaliplatin
- Capecitabine and Oxaliplatin (Active Comparator): Capecitabine and Oxaliplatin
  Interventions: Drug: Capecitabine & Oxaliplatin

INTERVENTIONS:
Drug: S-1 & Oxaliplatin — S-1 and Oxaliplatin : S-1 80 mg/m2/day, D1-14 Oxaliplatin, 130 mg/m2/day, D1 Repeated every 3 weeks
  Other Names: S-1 and Oxaliplatin
  Arms: S-1 and Oxaliplatin
Drug: Capecitabine & Oxaliplatin — COX : Capecitabine 1000 mg/m2/day, D1-14 Oxaliplatin, 130 mg/m2/day, D1 Repeated every 3 weeks
  Other Names: Capecitabine and Oxaliplatin
  Arms: Capecitabine and Oxaliplatin

SUMMARY:
Primary objective :

To compare the combination of S-1 and oxaliplatin(SOX) to the combination of capecitabine and oxaliplatin(COX) therapy for advanced or metastatic colorectal carcinoma.

Secondary objectives :

1. To evaluate and compare the efficacy (overall survival and response rate) in the two treatment groups.
2. To evaluate and compare the quality of life of the patients and safety profiles of the two treatment groups.

DETAILED DESCRIPTION:
* The urgent need for new effective therapy with better safety profile for metastatic colorectal cancer patients and promising results observed so far in trials with S-1 combined with oxaliplatin in gastrointestinal cancer including colorectal cancer strongly warrants the comparison of S-1 combined with oxaliplatin to capecitabine combination with oxaliplatin acknowledged as a standard regimen in a first-line treatment for advanced colorectal cancer patients.
* Recently, a Phase I study was completed, indicating recommended dose as S-1 100 mg/m2/day1-14 and oxaliplatin (130 mg/m2/day1), repeated every 3 weeks. However, in the phase II study using the above recommended dose, delayed toxicities of thrombocytopenia and anemia were observed. These delayed toxicities were also reported in a phase II study using S-1 90 mg/m2/day plus oxaliplatin 130 mg/m2/day1 in advanced gastric cancer. At 2007 GI ASCO, the interim data of S-1(80 mg/m2/day1-14) plus oxaliplatin (130 mg/m2/day1) combination, repeated every 3 weeks, was presented, showing promising antitumor activity with favourable safety profile. Among 18 patients, there were only two patients with Grade 3 thrombocytopenia and one with Grade 3 neutropenia. Response rate was 57.1 % and disease control rate was 92.9 %. Considering these results and Japanese data which showed that enhanced efficacy was not observed with S-1 over 90 mg/m2/day and oxaliplatin combination, S-1 80 mg/m2/day 1-14 and oxaliplatin 130 mg/m2/D1, repeated every 3 weeks, will be tested in this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented colorectal adenocarcinoma
* Age over 18 years old
* Performance status (ECOG scale): 0-2
* Measurable or evaluable disease
* Patients can take food and drugs orally
* Adequate organ functions
* Life expectancy ≥ 3 months
* Patients should sign a written informed consent before study entry

Exclusion Criteria:

* Tumor type other than adenocarcinoma
* Second primary malignancy
* Prior systemic therapy (for instance, cytotoxic chemotherapy or active/passive immunotherapy) for advanced or metastatic colorectal cancer
* Adjuvant or neo-adjuvant treatment for non-metastatic (M0) disease has been completed within 6 months prior to initiation of study treatment.
* Prior radiotherapy was administered to target lesions selected for this study, or radiotherapy to the non-target lesions has been completed within 4 weeks before randomization.
* Presence of CNS metastasis
* Obvious peritoneal seeding or bowel obstruction disturbing oral intake
* Symptomatic peripheral neuropathy
* Major surgery within 4 weeks prior to study treatment start, or lack of complete recovery from the effects of major surgery. The patient received curative operation or RFA for metastatic disease.
* Serious illness or medical conditions
* Receiving a concomitant treatment with drugs interacting with S-1, capecitabine or oxaliplatin, as follows;flucytosine, a fluorinated pyrimidine antifungal agent phenytoin warfarin etc.
* Received any investigational drug or agent/procedure, i.e. participation in another trial within 4 weeks before beginning treatment with study drug.
* Pregnant or lactating woman
* Women of child bearing potential not using a contraceptive method
* Sexually active fertile men not using effective birth control during medication of study drug and up to 6 months after completion of study drug if their partners are women of child-bearing potential
* Any patients judged by the investigator to be unfit to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To compare the combination of S-1 and oxaliplatin to the combination of capecitabine and oxaliplatin in terms of progression free survival in patients previously untreated by systemic therapy for advanced or metastatic colorectal carcinoma. | 9 months

SECONDARY OUTCOMES:
To evaluate and compare the efficacy (overall survival and response rate) in the two treatment groups. | 24 months
To evaluate and compare the quality of life of the patients and safety profiles of the two treatment groups. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Young Suk Park, M.D.,Ph.D., Study Chair — Samsung Medical Center, Seoul, Korea; Hye Jin Kang, M.D.,Ph.D., Principal Investigator — Korea Cancer Center Hospital , Seoul, Korea; Jee Hyun Kim, M.D.,Ph.D., Principal Investigator — Seoul National University Bundang Hospital, Gyeonggi, Korea; Tae Won Kim, M.D.,Ph.D., Principal Investigator — Asan Medical Center, Seoul, Korea; Tae-Yoo Kim, M.D.,Ph.D., Principal Investigator — Seoul National University Hospital , Seoul, Korea; Dong Bok Shin, M.D.,Ph.D., Principal Investigator — Gil Medical Center, Gyeonggi, Korea; Joong Bae Ahn, M.D.,Ph.D., Principal Investigator — Yonsei Medical Center, Severance Hospital, Seoul, Korea; Kyung Hee Lee, M.D.,Ph.D., Principal Investigator — Yeungnam University College of Medicine , Daegu, Korea; Namsu Lee, M.D.,Ph.D., Principal Investigator — Soon Chun Hyang University Hospital , Seoul, Korea; Ik-Joo Chung, M.D.,Ph.D., Principal Investigator — Chonnam National University Hwasun Hospital, Jeollanamdo, Korea; Yong Sang Hong, M.D.,Ph.D., Principal Investigator — National Cancer Center, Gyeonggi, Korea
Locations (11):
- South Korea (11):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonnam National University Hospital, Hwasun, Jeollanamdo
  - Yeungnam University, Daegu
  - Gachon University Gil Medical Center, Inchon
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Korea Cancer Center Hospital, Seoul
  - Soon Chun Hyang University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University, Seoul

REFERENCES:
- [Derived] Kim ST, Hong YS, Lim HY, Lee J, Kim TW, Kim KP, Kim SY, Baek JY, Kim JH, Lee KW, Chung IJ, Cho SH, Lee KH, Shin SJ, Kang HJ, Shin DB, Lee JW, Jo SJ, Park YS. S-1 plus oxaliplatin versus capecitabine plus oxaliplatin for the first-line treatment of patients with metastatic colorectal cancer: updated results from a phase 3 trial. BMC Cancer. 2014 Nov 26;14:883. doi: 10.1186/1471-2407-14-883. PMID 25424120
- [Derived] Hong YS, Park YS, Lim HY, Lee J, Kim TW, Kim KP, Kim SY, Baek JY, Kim JH, Lee KW, Chung IJ, Cho SH, Lee KH, Shin SJ, Kang HJ, Shin DB, Jo SJ, Lee JW. S-1 plus oxaliplatin versus capecitabine plus oxaliplatin for first-line treatment of patients with metastatic colorectal cancer: a randomised, non-inferiority phase 3 trial. Lancet Oncol. 2012 Nov;13(11):1125-32. doi: 10.1016/S1470-2045(12)70363-7. Epub 2012 Oct 10. PMID 23062232